CLINICAL TRIAL: NCT05615597
Title: Evaluating the Efficacy of Para-discal Infiltration in Patients With Lateralized MODIC 1 Inflammatory Disc Disease: Pilot Study (IPAD)
Brief Title: Evaluating the Efficacy of Para-discal Infiltration in Patients With Lateralized MODIC 1 Inflammatory Disc Disease
Acronym: IPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL22_0230
Record Dates: First submitted 2022-10-27; First posted 2022-11-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Degenerative Disc Disease; Inflammation; Low Back Pain
Keywords: Low back pain; Injections; Degenerative Disc Disease; Inflammation
MeSH Terms: conditions — Intervertebral Disc Degeneration; Inflammation; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Para-discal infiltration (Other): Single arm study
  Interventions: Procedure: Para-discal injection of corticoid

INTERVENTIONS:
Procedure: Para-discal injection of corticoid — In this pilot study, all patients underwent the same procedure: a corticosteroid infiltration via a para-discal approach. The infiltrations were performed under CT or scopy.

SUMMARY:
Degenerative disc disease (DDD) is a major cause of chronic low back pain (> 40%). It can be defined by specific magnetic resonance imaging (MRI) features, with a strong correlation between pain and the inflammatory aspect of the disc, resulting in active disc disease (AD). The Modic classification based on MRI of the lumbar spine is considered a reference.

The management of low back pain in patients with inflammatory disc disease generally involves intra-disc corticosteroid infiltration, which has been widely proven to be effective in reducing pain [4-6]. However, this procedure can be painful and invasive and sometimes impossible to perform due to severe disc impingement.

The aim of this study is to evaluate the efficacy on pain of para-disc infiltration of corticosteroids in contact with the inflammatory MRI signal abnormality (Modic 1) when it is lateralized.

This variant of infiltration is easier to perform (no catheterisation of the disc and therefore quicker), would entail less risk of disc infection and would be accessible to more radiologists.

It is already practised but, to our knowledge, has never been the subject of a study to evaluate its effectiveness on pain.

If successful, more patients could be treated and the range of treatment could be extended.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient with Modic I lateralized disc disease seen on an MRI less than 6 months old.
* Chronic medial or lateralized (same side as MODIC 1) low back pain for at least 3 months with a mean pain intensity ≥ 40/100 mm on a VAS.
* Effective contraception for women of childbearing age, at least 6 months after injection (surgical sterilisation, approved hormonal contraceptives, barrier methods, intrauterine intrauterine device)

Exclusion Criteria:

* Patient with MODIC 1 in both underlying and overlying vertebral spaces.
* Patient with an inflammatory signal abnormality of the vertebral body plateau related to non-mechanical pathology (e.g. spondyloarthritis).
* Patients with a history of lumbar spine surgery.
* Patient with suspected spondylodiscitis or other infection.
* Patients on anticoagulant or antiaggregant therapy, or with a coagulation disorder.
* Patients with an allergy to iodine or to any of the components of Xylocaine.
* Patients with an allergy to prednisolone or to any component of Hydrocortancyl® or Dexamethasone®..
* Patient with severe uncontrolled disease (i.e. cardiac gastrointestinal, neurological, endocrine, autoimmune) that limits patient safety (as determined by the safety (as judged by the investigator).
* Prior to the treatment visit :

  * current and recent morphine use (< 1 month)
  * recent systemic or local corticosteroid therapy (< 1 month).
* Patient with sphincter disturbances indicative of cauda equina syndrome.
* Psychotic state not controlled by treatment
* Pregnancy (βHCG positive), breastfeeding
* Vulnerable patient protected by law
* Patient under guardianship or curatorship
* Patient participating in an interventional study
* Patient unable to read and/or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2025-07-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline pain using the Visual Analogue Scale (VAS) at 1 month | 1 month after intervention
  VAS pain is a subjective but simple and reproducible criterion and one of the most widely used to evaluate the effectiveness of a therapeutic strategy in chronic low back pain.
  0 represents no pain and 100 represents the worst pain imaginable.

SECONDARY OUTCOMES:
Concomitant treatments (analgesics/NSAIDs) | up to 6 months
  he use of analgesics or NSAIDs will be recorded throughout the study by direct questioning of the patient and/or through their medical records.
Change from The Oswestry Disability Index (ODI) at 1 month | 1 month after intervention
  The Oswestry Disability Index (ODI) is a validated questionnaire (Fairbank and Pynsent 2000). We will consider a patient as responder if he/she manages to achieve at least 30% improvement in ODI score between baseline and 1 month. This percentage of minimal improvement (30%) was judged to be a clinically relevant threshold by an international consensus conference (Ostelo et al. 2008).
Change from Baseline Pain using the Visual Analogue Scale (VAS) at 7 days | 7 days after intervention
  VAS pain is a subjective but simple and reproducible criterion and one of the most widely used to evaluate the effectiveness of a therapeutic strategy in chronic low back pain.
  0 represents no pain and 100 represents the worst pain imaginable.
Change from Baseline Pain using the Visual Analogue Scale (VAS) at 3 months | 3 months after intervention
  VAS pain is a subjective but simple and reproducible criterion and one of the most widely used to evaluate the effectiveness of a therapeutic strategy in chronic low back pain.
  0 represents no pain and 100 represents the worst pain imaginable.
Change from Baseline Pain using the Visual Analogue Scale (VAS) at 6 months | 6 months after intervention
  VAS pain is a subjective but simple and reproducible criterion and one of the most widely used to evaluate the effectiveness of a therapeutic strategy in chronic low back pain.
  0 represents no pain and 100 represents the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur HAMEL-SENECAL, MD, Principal Investigator — Departement of Medical Imaging - Montpellier University hospital LAPEYRONIE Hospital
Locations (1):
- Departement of Medical Imaging, Montpellier, Occitanie, France